CLINICAL TRIAL: NCT00918489
Title: A Phase II Study to Investigate the Efficacy and Tolerability of Vorinostat in Patients Suffering From Advanced, Metastatic Soft Tissue Sarcoma
Brief Title: Study on Efficacy and Tolerability of Vorinostat in Patients With Advanced, Metastatic Soft Tissue Sarcoma (STS)
Acronym: SAHA-I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gerlinde Egerer, Prof. Dr. med., Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHA-I
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Soft Tissue Sarcoma
Keywords: soft tissue sarcoma; metastatic; vorinostat
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat (Experimental): Daily administration of 400mg vorinostat on 28 days (one therapy cycle). Seven days of therapy break between two consecutive cycles.
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Daily administration of 400mg vorinostat on 28 days (one therapy cycle). Seven days of therapy break between two consecutive cycles.

SUMMARY:
Primary objective of the study is to investigate the efficacy of vorinostat in patients suffering from selected histological types of soft tissue sarcoma. Further evaluations relate to the safety and tolerability of vorinostat, its pharmacokinetics (course of plasma concentration over time) and pharmacodynamics (mode of action). Only subjects with advanced, metastatic disease will be included in this trail.

DETAILED DESCRIPTION:
The treatment with vorinostat will be administered daily over 28 days. This period will be referred to as a therapy cycle. Two consecutive therapy cycles will be separated by a 7-days therapy break. In case of a good response and no relevant side effects, the treatment with vorinostat can be continued for up to 1 year after begin of the treatment. If any relevant side effects or intolerability occur, the dose and/or schedule of administration will be modified according to the pre-defined criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with verified, metastatic soft tissue sarcoma of the following histologies:

   * undifferentiated highgrade pleomorphic sarcoma/pleomorphic malignant fibrous histiocytoma,
   * undifferentiated pleomorphic sarcoma with grand cells/grand cell fibrotic histiocytoma,
   * undifferentiated pleomorphic sarcoma with prominent inflammation/inflamed MFH,
   * myxofibrosarcoma,
   * liposarcoma,
   * synovial sarcoma,
   * rhabdomyosarcoma (pleomorph, alveolar und embryonal),
   * leiomyosarcoma,
   * adult fibrosarcoma,
   * angiosarcoma,
   * malignant hemangiopericytoma/ malignant solitaire fibrous tumor,
   * malignant peripheral neurilemma tumor,
   * extraskeletal mesenchymal chondrosarcoma,
   * extraskeletal myxoid chondrosarcoma,
   * undifferentiated sarcoma of non other specified (NOS) type.
2. Verified relapse or disease progression at study inclusion, i.e. therapeutic failure of the first line therapy with anthracyclines,
3. Measurable disease according to the RECIST criteria,
4. Previous systemic therapy of advanced and/or metastatic disease,
5. An interval of at least 4 weeks since the last surgery, chemotherapy or radiation,
6. Age over 18,
7. Following laboratory findings:

   * ANC ≥ 1.0 x 10³/mm³,
   * platelets ≥ 100.000/mm³,
   * hemoglobin ≥ 9 g/dl,
   * creatinin < 1.5 x ULN (upper limit of normal),
   * AST and ALT < 2.5 x ULN,
   * total bilirubin < 1.5 x ULN,
8. Life expectancy of at least 12 weeks,
9. Negative pregnancy test,
10. Consent for an effective contraception during and up to 6 month after the study completion.
11. Written informed consent,
12. Ability to understand the goal and the consequences of this trial.

Exclusion Criteria:

1. Proof of the following histologies:

   * gastrointestinal stromal tumor (GIST),
   * malignant mesothelioma,
   * neuroblastoma,
   * osteosarcoma,
   * Ewing's sarcoma/PNET,
2. Concurrent radio- or chemotherapy,
3. Participation in another interventional trial within 4 weeks prior to the inclusion,
4. Previous therapy with another HDAC-inhibitor (e.g. depsipeptide, MS-275, LAQ-824, PXD-101 und valproic acid). Patients, who underwent a therapy with valproic acid for treatment of seizures, can be included after a wash-out period of at least 30 days,
5. Symptomatic brain metastases, that have not been treated by radiotherapy. The interval between the last radiation and the study inclusion must not be shorter than 30 days,
6. Previous malignant disease (except for a non-melanoma of the skin and a carcinoma in situ of uterus), unless in complete remission and after the last therapy for at least 5 years,
7. Ejection fraction < 40 %,
8. Nursing,
9. Known allergy against the IMP or drugs with similar chemical structure or additives,
10. Active hepatitis B and/or C and HIV-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of vorinostat on the basis of progression free survival (PFS) up to 1 year after first administration of the IMP. | Up to 1 year

SECONDARY OUTCOMES:
Evaluation of the efficacy of vorinostat on the basis of overall survival up to 1 year after first administration of the IMP. Investigation on pharmacokinetics und pharmacodynamics of vorinostat. Evaluation of safety and tolerability of vorinostat. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gerlinde Egerer, MD, Study Director — Department of Internal Medicine V, Universtity Hospital Heidelberg
Locations (7):
- Germany (7):
  - Department of Hematology, Oncology, Rheumatology and Immunology, University Hospital Tübingen, Tübingen, Baden-Wurttemberg
  - Department of Hematology, Hemostaseology, Oncology and Stemm Cell Transplantation, Medical School Hannover, Hanover, Niedersachen
  - Department of Oncology, Hematology and Palliative Medicine, Marien Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Comprehensive Cancer Center North, University Hospital Kiel, Kiel
  - Sarcoma Center Mannheim, University Hospital Mannheim, Mannheim
  - Center for Soft Tissue Sarcoma, University Hospital Tübingen, Tübingen
  - Comprehensive Cancer Center Ulm (CCCU), Ulm

REFERENCES:
- [Derived] Schmitt T, Mayer-Steinacker R, Mayer F, Grunwald V, Schutte J, Hartmann JT, Kasper B, Husing J, Hajda J, Ottawa G, Mechtersheimer G, Mikus G, Burhenne J, Lehmann L, Heilig CE, Ho AD, Egerer G. Vorinostat in refractory soft tissue sarcomas - Results of a multi-centre phase II trial of the German Soft Tissue Sarcoma and Bone Tumour Working Group (AIO). Eur J Cancer. 2016 Sep;64:74-82. doi: 10.1016/j.ejca.2016.05.018. Epub 2016 Jun 28. PMID 27367154